CLINICAL TRIAL: NCT06673030
Title: Evaluation of the Effectiveness of Kaleidoscope and Tell-Show-Play-Doh in Reducing Dental Anxiety for Children Undergoing Pulpotomy in Primary Molars - a Randomized Controlled Clinical Trial
Brief Title: Evaluation of the Effectiveness of New Management Techniques in Reducing Dental Anxiety for Children Undergoing Pulpotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Eman Mohamed Yousef Mohamed Elmansy, Master's degree student, Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Mansoura University, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A01011023PP
Record Dates: First submitted 2024-10-29; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Anxiety
Keywords: Childhood dental anxiety, Behavior management.
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Tell-Show-Do) (Active Comparator)
  Interventions: Other: Group 1 (Tell-Show-Do)
- Group 2 ( Tell-Show-Play-Doh) (Experimental)
  Interventions: Behavioral: The Play-Doh Doctor Drill 'n Fill toy set
- Group 3 (Kaleidoscope glasses ) (Experimental)
  Interventions: Behavioral: Using Kaleidoscope glasses during pulpotomy procedures

INTERVENTIONS:
Behavioral: Using Kaleidoscope glasses during pulpotomy procedures — Kaleidoscope is an instrument that shows an infinite number of fascinating geometric shapes in the form of a flower, repeating and reflecting images of coloured goggle fragments in the front section in a prism mirroring the inner surface.
  Arms: Group 3 (Kaleidoscope glasses )
Behavioral: The Play-Doh Doctor Drill 'n Fill toy set — Consists of a plastic human head with slots into which Play-doh molded teeth can be inserted. A battery operated toy drill is used to drill into and clean the black, cavitated tooth model and filled with white Play-Doh compound to simulate cavity preparation and restoration using tooth colored cement.
  Arms: Group 2 ( Tell-Show-Play-Doh)
Other: Group 1 (Tell-Show-Do) — In which Tell-Show-Do technique was done in three stages:
  * Tell: The dental procedures were explained to the children using language and expressions appropriate for their age.
  * Show: This began with showing the child the instruments and the topical anesthetic gel, high-speed handpiece and explaining the purpose of using the handpiece. and how the water removed using the suction device.
  * Do: Performing the dental procedure immediately.
  Arms: Group 1 (Tell-Show-Do)

SUMMARY:
The goal of this clinical trial is to reduce dental anxiety for sixety six children undergoing pulpotomy in primary molars by using kaleidoscope glasses and Tell-Show-Play-Doh techniques and evaluation of behavior and anxiety achieved by using FLAAC scale, measuring heart rate and RMS-Pictorial scale.

ELIGIBILITY:
Inclusion Criteria: 1. Children attended the dental clinic for their first time.

2. Children aged between 4 to 6 years including both boys and girls. 3. Healthy Children with Frankl's behavior rating score 2,3 and 4 of Frankl's behavior rating scale and no prior dental experience.

4. Children with carious lesions in lower restorable primary molars and indicated for pulpotomy.

- Exclusion Criteria: 1.Children with known significant visual impairments or psychological problems.

2. Children suffering from systemic diseases or special health care needs.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2023-08-05 (Actual); Primary Completion 2024-03-09 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Assessment of behavior of the child before and during and after the pulpotomy procedures. | Pre-operatively , during the procedure and post-operatively at the end of the visit at the same visit with no follow up.
  * Assessment of behavior of the child using ( Frankl's behavior rating scale to measure the cooperation behavior of the child, FLACC scale ).
  * Frankl's behavior rating scale was used pre-operatively and post-operatively with 4 scores : score 1(Definitely negative) score 2(Negative) score 3(Positive) score 4 (Definitely positive), the best scores for positive attitude and cooperation are score 3, 4.
  * The FLACC scale was used to measure behavior of the child according to Face, Legs, Activity, Cry and Consolability during the pulpotomy procedures with Scores: (0 = Relaxed and comfortable) (1-3 = Mild discomfort ) (4-6 = Moderate pain) (7-10 = Severe discomfort/pain).
Assessment of anxiety of the child before and after the pulpotomy procedures. | Pre-operatively and post-operatively at the end of the visit at the same visit with no follow up.
  * Assessment of anxiety of the child using (Pulse Oximeter to measure heart rate pre-operatively and post-operatively, RMS Pictorial Scale at the end of the visit). Increasing in heart rate readings means increasing anxiety.
  * RMS Pictorial Scale which comprises a row of five faces ranging from score 1(very happy) to score 5 (very unhappy) and the children were asked to choose the face they felt like about themselves at that moment.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Mansoura university, Mansoura, Egypt., Egypt

IPD SHARING:
Plan to Share IPD: No